CLINICAL TRIAL: NCT02801357
Title: A Phase 1 Study to Evaluate the Relative Exposures of Lofexidine and Its Major Metabolites in Subjects Seeking Buprenorphine Dose Reduction
Brief Title: Study to Evaluate the Exposures of Lofexidine and Its Major Metabolites in Subjects Seeking Buprenorphine Dose Reduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM- LX1-1013
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Substance Withdrawal Syndrome; Opiate Addiction; Opiate Dependence
Keywords: substance withdrawal syndrome; opiate addiction; opiate dependence; opioid withdrawal syndrome; buprenorphine
MeSH Terms: conditions — Substance Withdrawal Syndrome; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lofexidine with tapering buprenorphine (Experimental): Enrolled subjects must be on a daily dose of between 8 - 24 mg of buprenorphine for at least 30 days. Once enrolled, subjects will receive lofexidine as follows: Days 1 through 3, 0.6 mg 4 times daily (QID; 2.4 mg daily); Days 4 through 6, 0.8 mg QID (3.2 mg daily), and Day 7 0.8 mg at 8 AM. Subjects will take their scheduled lofexidine doses at approximately 8 AM, 1 PM, 6 PM and 11 PM. Subjects will also reduce their current buprenorphine dose by at least 4 mg on Day 1.
  Interventions: Drug: lofexidine administration in subjects seeking buprenorphine dose reduction

INTERVENTIONS:
Drug: lofexidine administration in subjects seeking buprenorphine dose reduction

SUMMARY:
The purpose of this study is to evaluate the relative exposures of lofexidine and its major metabolites in subjects seeking buprenorphine dose reduction.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, inpatient study in male and female subjects seeking at least a 4 mg reduction of their buprenorphine maintenance dose. The purpose of this study is to assess the relative exposures of lofexidine and its 3 major metabolites in subjects tapering from buprenorphine maintenance treatment. Lofexidine is an alpha-2 adrenergic agonist under development for the treatment of acute withdrawal from short-acting opioids.

ELIGIBILITY:
Inclusion Criteria:

* Have current dependency such that the subject is maintained on a daily dose between 8 and 24 mg of buprenorphine and is seeking reduction of their buprenorphine dose by at least 4 mg.
* Urine toxicology screen positive for buprenorphine at Screening.
* Agree to collection of blood samples for genotyping of CYP2D6 metabolizer status.
* If female and of childbearing potential, subject must have been using birth control for at least 30 days and must agree to use an acceptable form of birth control through at least 30 days after the last dose of study drug.
* If male, must agree to use an acceptable form of birth control throughout the entire study period and for 90 days after the last dose of study drug. Must not donate sperm for 90 days after the last dose of study drug.

Exclusion Criteria:

* Be a female subject who is pregnant or lactating.
* Have a very serious medical illness not under control.
* Have participated in an investigational drug study within the past 30 days.
* Received any drugs that are known strong, moderate or weak inhibitors of cytochrome P450 (CYP) enzymes CYP1A2, CYP2C19, or CYP2D6, within 14 days or 5 half-lives (whichever is more) before Day -1.
* Abnormal cardiovascular exam at Screening.
* Subjects requiring the following will be excluded: Tricyclic antidepressants, which may reduce the efficacy of imidazoline derivatives; Beta-receptor blockers, to avoid the risk of excessive bradycardia.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Predose and peak metabolite (N-[2- aminoethyl-2-[2,6-dichlorophenoxy] propanamide [LADP], 2-[2,6-dichlorophenoxy] propionic acid [LDPA] and 2,6-Dichlorophenol [2,6-DCP]) plasma concentration to lofexidine (parent) ratios on each day of treatment | pre-1 PM dose and 3 hours post-1 PM dose on Days 1-6; pre-8 AM dose and 1, 3, 7, 12, 24, and 34 hours post-8 AM dose on Day 7

SECONDARY OUTCOMES:
Modified Clinical Global Impression - subject and observer | 3.5 hours post-8 AM dose on Days 1-7
Visual Analog Scale for Efficacy | 3.5 hours post-8 AM dose on Days 1-7
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline: Day -1; 3.5 hours post-first dose on Day 1; Day 8
Holter ECGs | Day -1; pre-1 PM dose, 3 and 4 hours post-1 PM dose on Days 1 and 6
Blood pressure and pulse (sitting and standing) | screening; Day -1; within 30 minutes before every dose Days 1-8
Laboratory Assessments | screening
  Measurements in hematology, chemistry, urinalysis, infectious disease panel. Labs will be done at screening.
Oral temperature and respiration | screening; Day -1; pre-8 AM dose on Days 1-8
12-Lead ECG | screening
Adverse Events Assessment | Day -1; Days 1-8
Urine drug screening | Screening; Day -1, Days 1-8
Concomitant medications | Screening; Day -1, Days 1-8
Physical exam | screening; Day -1; Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No